## **Cover Page**

Official title of the study: Coil Hysteroscopic Tubal Occlusion,

the Treatment of Hydrosalpinx Before IVF-ET

**Date:** 12/01/2015

## Statistical Analysis Plan

- 1. Measurements used: Successful placement of coils will be judged by the correct placement that confirmed by vaginal ultrasound examination. Implantation rate, first-trimester spontaneous miscarriage rate and on-going pregnancy rate will also be calculated.
- 2. Sample size calculation: As a single-arm trial, 80 females will be recruited in our study.
- 3. Statistical methods: Data analysis was performed with SPSS version 22.0 (SPSS, Inc., Chicago, IL, USA), using two-sided test, and a p value < 0.05 was considered statistically significant. The participants who received insertion of fibered coils were followed up and the outcomes were recorded. Chi-square test will be applied to evaluate the basic data of the participants including age and IVF-ET cycles. Ratio was applied in the outcomes of miscarriage rate and pregnancy rate.